CLINICAL TRIAL: NCT06069414
Title: Atelectasis Evaluated With Lung Ultrasound After Inhalation or Intravenous Induction in Pediatric Anesthesia: a Prospective, Observational, Propensity Scored Matched Study
Brief Title: Atelectasis After Inhalation or Intravenous Induction in Pediatric Anesthesia
Acronym: AtelectLUS
Status: Completed | Type: Observational
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Principal Investigator, Vittore Buzzi Children's Hospital
Other Study IDs: 2022/ST/147
Record Dates: First submitted 2023-09-13; First posted 2023-10-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Atelectasis; Pediatric Anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalatory induction: Patients who will be induced via mask with inhalators anesthetic gases
  Interventions: Other: Type of anesthesia induction
- Intravenous induction: Patients who will be induced with intravenous anesthetics
  Interventions: Other: Type of anesthesia induction

INTERVENTIONS:
Other: Type of anesthesia induction — Patients will receive inhalatory or intravenous anesthesia at their choice; both groups will be evaluated with lung ultrasound after induction to detect ultrasonografic signs of atelectasis

SUMMARY:
Children have a highly compliant chest wall and atelectasis formation occurs often during pediatric anesthesia. Inhalation induction is commonly performed in pediatric anesthesia but it is still unclear if this can have an effect on the development of atelectasis. Aim of this study is to investigate the impact of inhalation versus intravenous induction on atelectasis formation during anesthesia induction in children. Atelectasis will be evaluated with lung ultrasound before induction and right after induction.

DETAILED DESCRIPTION:
Respiratory complications, among which atelectasis, are a common cause of adverse events in pediatric anesthesia. Lung ultrasound (LUS) examination is a point of care, non-invasive, radiation-free tool with high sensitivity and specificity for the identification of anesthesia-induced atelectasis in children.

Inhalation induction is commonly performed in pediatric anesthesia to avoid pain at venipuncture or to facilitate vein cannulation. This technique has been associated with a higher rate of respiratory adverse events but no study has investigated the role of inhalation or intravenous induction on lung atelectasis development in pediatric anesthesia.

The investigators will perform this study aiming to describe the impact of inhalation versus intravenous induction technique on atelectasis formation during anesthesia induction in children of different ages.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery under general anesthesia
* parental consent

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status III-VI
* neuromuscular disease
* chronic lung disease
* cardiopathy
* thoracic cage malformations
* chronic home ventilation (either invasive or non-invasive)
* positive history of foreign body inhalation
* required immediate life-saving procedures
* lack of parental consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 years of age scheduled for general anesthesia due to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Global LUS score | Upon completion of induction and subsequent controls at end of surgery and 1 postoperative day
  Sum of the LUS scores given to all the lung areas. Score points vary from 0 to 3, where 0 means normality of the lung and 3 refers to complete loss of aeration-tissue-like pattern or consolidation.
Signs of atelectasis | Upon completion of induction and and subsequent controls at end of surgery and 1 postoperative day
  Number of lung areas presenting a sub pleural consolidation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Camporesi, M.D., Study Director — Vittore Buzzi Children's Hospital
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sargent MA, McEachern AM, Jamieson DH, Kahwaji R. Atelectasis on pediatric chest CT: comparison of sedation techniques. Pediatr Radiol. 1999 Jul;29(7):509-13. doi: 10.1007/s002470050632. PMID 10398785
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Zeng C, Lagier D, Lee JW, Vidal Melo MF. Perioperative Pulmonary Atelectasis: Part I. Biology and Mechanisms. Anesthesiology. 2022 Jan 1;136(1):181-205. doi: 10.1097/ALN.0000000000003943. PMID 34499087
- [Background] Adler AC, Siddiqui A, Chandrakantan A, Matava CT. Lung and airway ultrasound in pediatric anesthesia. Paediatr Anaesth. 2022 Feb;32(2):202-208. doi: 10.1111/pan.14337. Epub 2021 Dec 1. PMID 34797019
- [Result] de Graaff JC, Bijker JB, Kappen TH, van Wolfswinkel L, Zuithoff NP, Kalkman CJ. Incidence of intraoperative hypoxemia in children in relation to age. Anesth Analg. 2013 Jul;117(1):169-75. doi: 10.1213/ANE.0b013e31829332b5. Epub 2013 May 17. PMID 23687233
- [Derived] Camporesi A, Roveri G, Vetrugno L, Buonsenso D, De Giorgis V, Costanzo S, Pierucci UM, Pelizzo G. Lung ultrasound assessment of atelectasis following different anesthesia induction techniques in pediatric patients: a propensity score-matched, observational study. J Anesth Analg Crit Care. 2024 Oct 5;4(1):69. doi: 10.1186/s44158-024-00206-x. PMID 39369249